CLINICAL TRIAL: NCT03872063
Title: Efficacy of a Physiotherapy Program Through Myofascial Induction and Eccentric Exercises in the Improvement of Mobility and the Perception of Nonspecific Pain in the Shoulder Joint in Volleyball Players. A Randomized Pilot Study
Brief Title: Myofascial Induction and Eccentric Exercises in Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RADO
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Myofascial Pain
Keywords: Volleyball; Range of motion; Myofascial; Eccentric; Pain
MeSH Terms: conditions — Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial (Experimental): Each session will last 17 minutes, taking place for 1 day a week, in a period of 4 weeks. The intervention will be carried out at the end of the training session. After the training, the technique of myofascial induction and eccentric exercises will be performed.
  Interventions: Other: Experimental
- Eccentric (Active Comparator): Each session will have a duration of 9 minutes, taking place during 1 day a week, in a period of 4 weeks. The intervention will be carried out at the end of the training session. After the training, the eccentric exercises will be performed.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The intervention by myofascial induction will consist of the application of two techniques: global technique of myofascial induction of the pectoralis major muscle (once the tissue is placed in tension, the direction of fascia release in that region should be followed and as a result of the release, the caudal hand can move to the pelvis in any direction, to the right or to the left) and telescopic technique for the upper extremity of the subject's dominant arm (gently tractioning the upper limb of the subject, making a slight external rotation, so slow and progressive). The subjects will then perform the eccentric exercises, which will also be done by control group subjects
  Other Names: Myofascial
  Arms: Myofascial
Other: Control — The intervention by eccentric exercises will consist of two exercises using an elastic band. In the supine position, with the elastic band on the contralateral side attached to a fixed body perpendicular to the subject's hand performing a slow and constant movement of external rotation against resistance in an approximately 45 degree arc; holding for 5 seconds and relaxing slowly (perform 3 sets of 12 repetitions). The second exercise, with the elbow in 90 degrees of flexion and a shoulder abduction also of 90 degrees, with the elastic band in front of the subject, executing a movement against resistance performing an external rotation.
  Other Names: Eccentric exercises
  Arms: Eccentric

SUMMARY:
Introduction. Myofascial therapy aims to improve fascial restrictions through the application of mechanical stimuli. The eccentric exercises involve the recruitment of fast fibers and help increase muscle volume.

Aim. Compare the effectiveness of myofascial induction intervention in the improvement of the range of motion of glenohumeral rotation and the pain perception, with respect to the use of eccentric exercises in volleyball players from 18 to 35 years of age.

Study design. Multicenter and single-blind randomized clinical study with follow-up period.

Methods. A random assignment of the 40 subjects recruited to the different study groups will be carried out: experimental (myofascial induction technique and eccentric exercises) and control (eccentric exercises). The intervention will last 4 weeks, with a weekly session of 17 and 7 minutes (in the experimental and control group, respectively). The dependent variables and measurement instruments will be: internal and external shoulder rotation (goniometry) and pain perception (visual analog scale). The Kolmogorov-Smirnov test will calculate the distribution of the sample, using parametric tests (t-student to calculate the difference of means between the evaluations in each group and ANOVA of repeated measures to calculate the intra- and intersubject effect) in case of normal.

Expected results. To improve the range of motion of glenohumeral joint global rotation and of the perception of pain of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Volleyball players
* Both gender
* Age range of 18 to 35 years
* Compete in a federated team in the Community of Madrid.

Exclusion Criteria:

* Have an injury to the osteoarticular complex of the shoulder at the time of the study or the previous 6 months
* Who are receiving a physiotherapy intervention at the time of the study or receiving analgesic drugs
* Not signed the informed consent document.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline range of motion of shoulder after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The measurement of the range of motion of shoulder will be made by means of a goniometric evaluation. The physiotherapist will be placed homolateral to the shoulder of the subject, being in the supine position with 90º shoulder abduction and 90º elbow flexion. While the goniometer will be positioned with the fulcrum in the olecranon, the fixed arm projected in the direction of the styloid process of the ulna and the movable arm follows the movement of the ulna. The range of normal mobility of the internal rotation of the shoulder is 0-100º and the external rotation of 0-80º (the total glenohumeral rotation range of 180º) if measured from the longitudinal axis of the arm. The unit of measurement is the degree, with a higher score indicating greater mobility of the shoulder joint.

SECONDARY OUTCOMES:
Change from baseline perception of pain of the coracoid process after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of the perception of pain of the coracoid process to palpation will be made with the Analog Visual Scale. The patient will be asked to indicate the pain that refers to the palpation in the region of the anterior aspect of the shoulder, in the area of the coracoid process. With this test the pain score of the subject will be measured, who will point in a straight line without dot marking between two extremes. The score range of this scale is 0-10, where 0 indicates no pain and 10 the maximum pain capable to endure.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain